CLINICAL TRIAL: NCT05638269
Title: A Multicentre Study on Features of the Gut Microbiota of Patients With Critical Chronic Diseases in China
Status: Recruiting | Type: Observational
Sponsor: Zhujiang Hospital (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Principal Investigator, Yan He, Professor, Zhujiang Hospital
Other Study IDs: CALM2101
Record Dates: First submitted 2022-09-26; First posted 2022-12-06 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Essential Hypertension; Liver Cancer; Nasopharyngeal Cancer; Pancreatic Cancer; Lung Cancer; Chronic Kidney Diseases; Acute Coronary Syndrome; Epilepsy; Gastric Cancer; Primary Aldosteronism; Subclinical hypothyroïdism
Keywords: cardiovascular disease; exctracoonic cancer; nervous system diseases; endocrine diseases; urological diseases; microbial dysbiosis
MeSH Terms: conditions — Essential Hypertension; Liver Neoplasms; Nasopharyngeal Neoplasms; Pancreatic Neoplasms; Lung Neoplasms; Renal Insufficiency, Chronic; Acute Coronary Syndrome; Epilepsy; Stomach Neoplasms; Hyperaldosteronism; Cardiovascular Diseases; Nervous System Diseases; Endocrine System Diseases; Urologic Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Feces, saliva, urine, serum, plasma and buffy coat
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- disease group: no intervention
  Interventions: Other: no intervention
- control group: no intervention
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — Observational studies, no intervention

SUMMARY:
The human gut microbiome has been associated with many health factors but variability between studies limits the exploration of effects between them. This study aims to systematically characterize the gut microbiota of various critical chronic diseases, compare the similarities and differences of the microbiome signatures linked to different regions and diseases, and further investigate their impacts on microbiota-based diagnostic models.

DETAILED DESCRIPTION:
Many studies demonstrate that microbial dysbiosis has been linked to many human pathologies. However, the current understanding of the identification of the disease-associated microbiome signatures remains limited, largely owing to the heterogeneity of microbial community structures which are shaped by the host. Undoubtedly, profiles of microbial biomarkers require validation in large, independent, population-based cohorts from different districts. Based on these, the investigator plan to organize a multicentric cross-sectional cohort, not only to systematically characterize the gut microbiota of various critical chronic diseases, such as liver cancer, gastric cancer, pancreatic cancer, lung cancer, nasopharyngeal cancer, hypertension, acute coronary syndrome, primary aldosteronism, epilepsy, chronic kidney disease, and subclinical hypothyroidism but also to compare the similarities and differences of the microbiome signatures linked to different regions and different diseases and to further investigate their impacts on microbiota-based diagnostic models. In this study, for each kind of disease, the investigators expect to recruit 500 patients with a confirmed diagnosis and 500 sex- and age-matched controls, to record their information related to demography, body measurement, lifestyle, diet, medication, diseases, and biochemistry, and to collect their feces, saliva, urine and blood samples.

ELIGIBILITY:
Inclusion Criteria:

1. aged 18-75 years;
2. living in the province where the hospital is located in the last three years;
3. with a medical diagnosis of one of the target diseases;
4. willing to provide written informed consent.

Exclusion Criteria:

1. female in pregnancy or lactation(unless the subject is pregnant women);
2. with medical diagnoses of other serious illnesses;
3. with a history of bariatric surgery or intestinal resection, except for appendectomy；
4. individual who was treated with drugs in the preceding 1 month, including antibiotics, metformin, statins, acid inhibitor, probiotics, and probiotics; individuals having consumed yogurt more than 3 times in the preceding 1 month; heavy drinkers who have consumed more than 4 taels of liquor or 1000ml of beer; frequent alcohol consumers who have drunk per week in the last month.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All the patients with essential Hypertension, liver cancer, nasopharyngeal cancer, pancreatic cancer, lung cancer, chronic kidney disease, acute coronary syndrome, epilepsy, gastric cancer, primary aldosteronism or subclinical hypothyroidism hospitalized in our participant hospitals will be eligible to be enrolled. Also, their age- and sex-matched controls making a physical examination in the same hospital will be eligible to be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 12000 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
microbiome | baseline
  The microbial composition of the stool and saliva samples was determined by 16S rRNA (ribosomal ribonucleic acid) gene sequencing analysis and metagenomics. Comparison of microbial abundance and diversity of healthy volunteers and patients with various diseases.

SECONDARY OUTCOMES:
biochemistry | baseline
  Comparison of serum markers of healthy volunteers and patients with various diseases.
metabonomics | baseline
  Comparison of metabolites of healthy volunteers and patients with various diseases.
proteomics | baseline
  Comparison of peptides of healthy volunteers and patients with various diseases using mass spectrometry.

CONTACTS AND LOCATIONS:
Overall Officials: Yan He, Study Chair — Zhujiang Hospital
Locations (50):
- China (50):
  - Emergency General Hospital, Chaoyang, Beijing Municipality
  - The People's Hospital Of Nanchuan Chongqing, Nanchuan, Chongqing Municipality
  - YongChuan hospital of Chongqing Medical Univeristy, Yongchuan, Chongqing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Fujian Provincial Hospital, Fuzhou, Fujian
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - Lanzhou University Second Hospital, Lanzhou, Gansu
  - The Sixth Affiliated Hospital of South China University of Technology (Foshan Nanhai District People's Hospital ), Foshan, Guangdong
  - The First Affiliated Hospital of Jinan University（Guangzhou Overseas Chinese Hospital ）, Guangzhou, Guangdong
  - The seventh Affiliated Hospital, Sun Yat-sen University, Shenzhen, Guangdong
  - Zhongshan City People's Hospital, Zhongshan, Guangdong
  - The Second Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - People's Hospital of Guangxi Zhuang Autonomous Region, Nanning, Guangxi
  - Wuzhou Red Cross Hospital, Tongliao, Guangxi
  - The Affiliated Cancer Hospital of Guizhou Medical University, Guiyang, Guizhou
  - The Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou
  - Hainan Traditional Chinese Medicine Hospital, Haikou, Hainan
  - Daqing People's Hospital（The Fifth Affiliated Hospital of Harbin Medical University）, Daqing, Heilongjiang
  - The First Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The Sixth Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Jixi Ji Mine Hospital, Jixi, Heilongjiang
  - Qiqihar Hospital of Traditional Chinese Medicine, Qiqihar, Heilongjiang
  - Luoyang Maternal and Child Health Hospital, Luoyang, Henan
  - Cancer Hospital, The First Affiliated Hospital, College of Clinical Medicine,Medical College of Henan University of Science and Technology, Luoyang, Henan
  - Shangqiu First People's Hospital, Shangqiu, Henan
  - Wuhan Mental Health Center, Wuhan, Hubei
  - Xiangyang Central Hospital, Xiangyang, Hubei
  - Nanzhang People's Hospital, Xianyang, Hubei
  - Zhuzhou Central Hospital, Zhuzhou, Hunan
  - Affiliated Hospital of Inner Mongolia Minzu University, Wuzhou, Inner Mongolia
  - Wuxi No.2 People's Hospital, Wuxi, Jiangsu
  - Affiliated Hospital of Jinggangshan University, Ji’an, Jiangxi
  - First Affiliated Hospital of Gannan Medical University, Ganzhou, Jiangx
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangx
  - Chang Zhi Yi Xue Yuan Fu Shu He Ji Yi Yuan, Changzhi, Shanxi
  - The Second Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - The Hospital of Shanxi University of Chinese Medicine, Taiyuan, Shanxi
  - Xi'an People's Hospital (Xi'an Fourth Hospital), Xi’an, Shanxi
  - The First Affiliated Hospital of Xi'an Medical University, Xi’an, Shanxi
  - The General Hospital of Western Theater Command PLA, Chengdu, Sichuan
  - Guang'an People's Hospital, Guang’an, Sichuan
  - The People's Hospital of Leshan, Leshan, Sichuan
  - Tianjin Binhai New Area Dagang Hospital, Binhai, Tianjin Municipality
  - Tianjing Medical University Cancer Institute & Hospital, Dayingmen, Tianjin Municipality
  - Tianjin Beichen Hospital, Guoyuan Xincun, Tianjin Municipality
  - The First People's Hospital of Kashgar Prefecture, Kashgar, Xinjiang Uygur Autonomous Region
  - First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - Qunjing Hospital of Traditional Chinese Medicine, Qujing, Yunnan
  - Hwa Mei Hospital,University of Chinese Academy of Sciences, Ningbo, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] He Y, Wu W, Zheng HM, Li P, McDonald D, Sheng HF, Chen MX, Chen ZH, Ji GY, Zheng ZD, Mujagond P, Chen XJ, Rong ZH, Chen P, Lyu LY, Wang X, Wu CB, Yu N, Xu YJ, Yin J, Raes J, Knight R, Ma WJ, Zhou HW. Regional variation limits applications of healthy gut microbiome reference ranges and disease models. Nat Med. 2018 Oct;24(10):1532-1535. doi: 10.1038/s41591-018-0164-x. Epub 2018 Aug 27. PMID 30150716